CLINICAL TRIAL: NCT02236247
Title: Heart Rate Control as an Additional Therapeutic Strategy in Patients With Decompensated Heart Failure: a Prospective, Randomized, Double-blinded, Placebo-controlled Study.
Brief Title: Control of Sinus Node Tachycardia as an Additional Therapy in Patients With Decompensated Heart Failure
Acronym: CONSTATHE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marco Stephan Lofrano Alves, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE:09145612.8.0000.0068; 2012/06163-6 (Other Grant/Funding Number: FAPESP - SAO PAULO RESEARCH FOUNDATION)
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Decompensated Heart Failure
Keywords: ivabradine; heart rate; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ivabradine (Experimental): I(f) inhibitor, heart rate controller
  Interventions: Drug: ivabradine
- placebo (Placebo Comparator): placebo pill will be administered orally twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ivabradine — 5 mg oral twice daily
  Other Names: procoralan
  Arms: ivabradine
Drug: Placebo — A placebo pill (identical to ivabradine) will be administered twice daily
  Arms: placebo

SUMMARY:
Study aims to compare the I(f) inhibitor ivabradine with placebo as strategy of heart rate control in patients with decompensated heart failure (DHF).

DETAILED DESCRIPTION:
Sympathetic hyperactivity and consequent increase in heart rate (HR) are physiological responses to low cardiac output in patients with decompensated heart failure (DHF). However, elevated HR may become inappropriate in these patients, increasing myocardial oxygen demand and decreasing diastolic filling time and might lead to hemodynamic deterioration, ventricular dysfunction (tachycardiomyopathy) and clinical deterioration.

Studies show the elevated HR is a predictor of poor prognosis in DHF. Subanalyses of large clinical trials using beta blockers (BBs) demonstrate the adequate control of HR correlates with a better outcome in patients with stable chronic heart failure (HF). However, use of BBs in patients with DHF is limited due to negative inotropic and hypotensive effects of these drugs.

As alternative to BBs, ivabradine has shown to increase survival of patients with chronic stable systolic HF. Compared to BBs, ivabradine has the advantage of "pure" negative chronotropic effect, no effect on myocardial contractility or peripheral vascular resistance. Despite the inhibition of I (f) has been validated as a therapeutic option in patients with stable HF, there are no studies available on this strategy in patients with DHF.

We hypothesized that HR control by ivabradine might improve clinical, hemodynamic and neurohormonal parameters in patients with DHF. The aim of this study was to evaluate the efficacy of HR control with ivabradine in patients with DHF.

ELIGIBILITY:
Inclusion Criteria:

* Sinus node rhythm
* HR> 80 bpm
* Hospitalization for DHF
* Ejection fraction ≤ 40%
* Sign informed consent

Exclusion Criteria:

* Systolic blood pressure <85 mmHg
* Signs of hypoperfusion
* Dobutamine>15 mcg/Kg/min
* Acute myocarditis
* Primary valvular disease requiring surgery
* Stroke in the last three months
* Hypertrophic or restrictive cardiomyopathy
* Sinus node disease
* Atrial fibrillation or flutter
* Second or third degree atrio-ventricular blockade
* Long QT syndrome
* Severe pulmonary disease
* Pulmonary embolism in the last three months
* Need for invasive ventilatory support
* Septicemia or septic shock
* Hepatic failure
* Creatinine > 2.5 mg/dL
* Hemodialysis
* Advanced malignancy
* Pregnancy or lactation
* Immunosuppressive therapy
* Use of cytochrome P450 inhibitors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline heart rate | Baseline, day 5 after intervention
  Heart rate will be assessed at morning, after 30 minutes of rest, recorded by electrocardiogram.

SECONDARY OUTCOMES:
Change from baseline blood pressure | Baseline, day 5 after intervention
  Blood pressure will be measured at morning by electronic cuff
Change from baseline ejection fraction | Baseline, day 5 after intervention
  Ejection fraction will be measured by echocardiography using Simpson´s rule
Change from baseline stroke volume | Baseline, day 5 after intervention
  Stroke volume will be measured by echocardiography using Doppler velocity-time integral technique.
Change from baseline creatinine | Baseline, day 5 after intervention
  Serum creatinine will be measured
Change from baseline brain natriuretic peptide | Baseline, day 5 after intervention
  Serum brain natriuretic peptide will be measured
Clinical | Up to 6 months
  Time of survival and free of readmission

OTHER OUTCOMES:
Safety/Adverse Event Outcome Measure | Up to day 15 days after intervention
  Number of Participants with Serious and Non-Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Edimar A Bocchi, MD-PHD, Study Chair — Heart Failure Unit, Heart Institute, University of Sao Paulo Medical School
Locations (1):
- Heart Failure Unit, Heart Institute, University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lofrano-Alves MS, Issa VS, Biselli B, Chizzola P, Ayub-Ferreira SM, Bocchi EA. Control of sinus tachycardia as an additional therapy in patients with decompensated heart failure (CONSTATHE-DHF): A randomized, double-blind, placebo-controlled trial. J Heart Lung Transplant. 2016 Oct;35(10):1260-1264. doi: 10.1016/j.healun.2016.06.005. Epub 2016 Jun 7. No abstract available. PMID 27469019
- See also: Related Info — http://www.jhltonline.org/article/S1053-2498(16)30172-3/abstract